CLINICAL TRIAL: NCT00868348
Title: Local Infiltration Analgesia for Total Knee Arthroplasty: Should Ketorolac be Added
Brief Title: A Comparison of Naropin and Ketorolac for Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-003180-39
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Pain
Keywords: Total Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Saline
- Ketorolac (Active Comparator)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — 30 mg (1 ml) infiltration combined with Intraarticular bolus injection of 120 mg (4 ml) ketorolac
  Other Names: Toradol
  Arms: Ketorolac
Drug: Saline — 1 ml infiltration 4 ml intraarticular bolus injection of placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to determine wether ketorolac is effective in the treatment of postoperative pain after total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty
* Age > 18
* Tolerance for study drugs
* Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjels Søballe, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University, Aarhus, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 361 patients were assessed for eligibility from May 2009 through March 2011; 62 patients participated in another study, 54 patients declined to participate, and 185 patients were excluded based on the exclusion criteria. Sixty patients (30 in each group)were enrolled, and data for the primary endpoint were registered in all patients
Groups:
- Control: Intraoperative local infiltration analgesia (ropivacaine 300 mg, epinephrine 0.5 mg and saline) After surgery,eight intra-articular bolus doses of ropivacaine 100 mg with saline
- Ketorolac: Intraoperative local infiltration analgesia (ropivacaine 300 mg, epinephrine 0.5 mg and ketorolac 30 mg) After surgery,eight intra-articular bolus doses of ropivacaine 100 mg with 15 mg ketorolac
Period: Overall Study
Arm/Group | Control | Ketorolac
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Gender, Age,
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 19 | 22 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [61 to 75] | 70 [65 to 75] | 71 [63 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  Denmark | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption
Description: Consumption of intravenous (i.v.) patient-controlled analgesia (PCA) morphine during the first forty-eight hours after surgery
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 30 | 30
mg | 48.75 [30 to 82.2] | 10 [0 to 22.5]

2. Secondary Outcome: Time to First i.v. Patient Controlled Analgesia (PCA) Morphine Request
Time Frame: within 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 30 | 30
min | 223 [115 to 319] | 490 [248 to 617]

3. Secondary Outcome: Pain Intensity Scores During Walking
Description: Pain intensity Visual Analogue Scale (VAS) (VAS; 0, no pain, and 100 mm, worst pain possible)
Time Frame: 6-24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 30 | 30
mm | 64 [51 to 80] | 29 [5 to 47]

4. Secondary Outcome: Home Readiness
Description: Ability to meet discharge criteria (home readiness)
Time Frame: time to fulfilment of discharge criteria
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 30 | 30
days | 3 [2 to 3] | 2 [2 to 3]

5. Secondary Outcome: Length of Hospital Stay
Time Frame: From the day of surgery until discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 30 | 30
days | 3 [3 to 3] | 3 [2 to 3]

6. Secondary Outcome: Pain Intensity During Daily Activity
Description: Pain intensity Visual Analogue Scale (VAS) (VAS; 0, no pain, and 100 mm, worst pain possible)
Time Frame: 16 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 28 | 29
mm | 4 [1 to 21] | 3 [3 to 12]

ADVERSE EVENTS:
Arm/Group | Control | Ketorolac
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=30) | Ketorolac (N=30)
Haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — re-admission due haematoma
tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Know tachycardia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes